CLINICAL TRIAL: NCT04841902
Title: Effects of Life Style Intervention Manual on Metabolic, Cardiovascular, Respiratory and Physical Parameters in Pre Hypertensive Sedentary Population
Brief Title: Effects of Life Style Intervention Manual in Pre Hypertensive Sedentary Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: REC/Lhr/21/1101 Danish Hassan
Record Dates: First submitted 2021-03-29; First posted 2021-04-12 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Pre Hypertension
Keywords: Pre Hypertension; Lifestyle Intervention; Metabolic parameters; Cardiovascular parameters; Respiratory parameters; Physical parameters
MeSH Terms: conditions — Prehypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Life Style Intervention Manual (Supervised) (Experimental): Supervised Exercises with Life Style Intervention Manual (Dietary & Educational Component) for 3 days / week for 16 weeks. Each session will comprise of 60 minutes of alternating light to moderate intensity aerobic exercises including warm up and rest interval
  Interventions: Other: Life Style Intervention Manual (With Exercise Under Supervision)
- Life Style Intervention Manual (Home Based) (Experimental): Home Based- Life Style Intervention Manual (Exercise, Dietary & Educational Component for 16 weeks. Subject will be asked to maintain a regular exercise and dietary diary to ensure adherence to the program
  Interventions: Other: Life Style Intervention Manual (Home Based)
- Control (Placebo Comparator): Age matched Control Group followed for 16 weeks with General Advise to stay healthy and active
  Interventions: Other: General Advice

INTERVENTIONS:
Other: Life Style Intervention Manual (With Exercise Under Supervision) — Life Style Intervention Manual for Pre Hypertensive subjects will consist of three components; Exercise, Dietary Modification and Education. The exercise will be supervised will other two components will be home based.
  Arms: Life Style Intervention Manual (Supervised)
Other: General Advice — General advice to stay healthy and active
  Arms: Control
Other: Life Style Intervention Manual (Home Based) — Life Style Intervention Manual for Pre Hypertensive subjects will consist of three components; Exercise, Dietary Modification and Education. All three components will be home based.
  Arms: Life Style Intervention Manual (Home Based)

SUMMARY:
Hypertension is an increasingly important medical and public health issue. The prevalence of hypertension increases with advancing age to the point where more than half of people 60-69 years of age and approximately three-fourths of those 70 years of age and older are affected. The age related rise in SBP is primarily responsible for an increase in both incidence and prevalence of hypertension with increasing age. At present, it is estimated that about 1 billion people worldwide have hypertension (>140/90 mmHg), and this number is expected to increase to 1.56 billion by 2025.

Because of the new data on lifetime risk of hypertension and the impressive increase in the risk of cardiovascular complications associated with levels of BP previously considered to be normal, the JNC 7 report has introduced a new classification that includes the term "prehypertension" for those with BPs ranging from 120-139 mmHg systolic and/or 80-89 mmHg diastolic. This new designation is intended to identify those individuals in whom early intervention by adoption of healthy lifestyles could reduce BP, decrease the rate of progression of BP to hypertensive levels with age, or prevent hypertension entirely. Prehypertension is not a disease category. Rather, it is a designation chosen to identify individuals at high risk of developing hypertension, so that both patients and clinicians are alerted to this risk and encouraged to intervene and prevent or delay the disease from developing. Individuals who are pre hypertensive are not candidates for drug therapy based on their level of BP and should be firmly and unambiguously advised to practice lifestyle modification in order to reduce their risk of developing hypertension in the future.

The goal for individuals with prehypertension and no compelling indications is to lower BP to normal levels with lifestyle changes, and prevent the progressive rise in BP using the recommended lifestyle modifications.

DETAILED DESCRIPTION:
Adoption of healthy lifestyles by all persons is critical for the prevention of high BP and is an indispensable part of the management of those with hypertension. Weight loss of as little as 10 lbs (4.5 kg) reduces BP and/or prevents hypertension in a large proportion of overweight persons, although the ideal is to maintain normal body weight. BP is also benefited by adoption of the Dietary approaches to Stop Hypertension (DASH) eating plan which is a diet rich in fruits, vegetables, and low fat dairy products with a reduced content of dietary cholesterol as well as saturated and total fat (modification of whole diet). It is rich in potassium and calcium content. Dietary sodium should be reduced to no more than 100 mmol per day (2.4 g of sodium). Everyone who is able should engage in regular aerobic physical activity such as brisk walking at least 30 minutes per day most days of the week. Lifestyle modifications reduce BP, prevent or delay the incidence of hypertension, enhance antihypertensive drug efficacy and decrease cardiovascular risk. For example, in some individuals, a 1,600 mg sodium DASH eating plan has BP effects similar to single drug therapy. Combinations of two (or more) lifestyle modifications can achieve even better results. For overall cardiovascular risk reduction, patients should be strongly counseled to quit smoking.

Lifestyle modification involves altering long-term habits, typically of eating or physical activity, and maintaining the new behavior for months or years. Lifestyle changes are a more natural way toward therapeutic goals and should be an integral component of halting or even reversing early vascular aging as in pre hypertensive subjects. From a public health perspective, even a small reduction in BP should have a tremendous, beneficial effect on the occurrence of hypertension and its complications. In view of the current epidemic of BP-related diseases and the proven effects of lifestyle modifications on BP, the current challenge to health care providers, researchers, and public officials is to develop and implement effective life style intervention program comprising exercise dietary and educative component in clinical and public health strategies that achieve and maintain healthy lifestyle modification

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 25 - 40 years
2. Either gender
3. Clinic BP will be consistent with the diagnosis of pre-hypertension
4. Sedentary Subjects (<150 min/week or <600 MET-min/week on IPAQ Urdu Version)

Exclusion Criteria:

1. Body Mass Index less than 18.5 kg/m2 or greater than 45 kg/m2
2. Evidence of target organ damage such as left ventricular hypertrophy, angina, heart failure, stroke, chronic kidney disease, peripheral artery disease
3. Women of child-bearing age who tested positive for HCG & breastfeeding women
4. Individuals who could not read the consent or Participated in another study within 3 months

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Blood Pressure | 16 Weeks
  Office, Ambulatory, Daytime, Nighttime & 24 hours Systolic & Diastolic Blood Pressure, Mean Arterial Blood Pressure measured at baseline, 8th Week post treatment and 16th Week post treatment
Change in Serum Triglycerides | 16 Weeks
  Serum Triglycerides measured at baseline, 8th Week post treatment and 16th Week post treatment
Change in Body Mass Index (BMI) | 16 Weeks
  Body Mass Index (BMI) measured at baseline, 8th Week post treatment and 16th Week post treatment. BMI is calculated using height (m) and weight (kg) using the formula kg/m^2
Change in Forced Vital Capacity (FVC) | 16 Weeks
  Forced Vital Capacity (FVC) measured at baseline, 8th Week post treatment and 16th Week post treatment using a digital spirometer.
Change in Serum Total Cholesterol | 16 Weeks
  Serum Total Cholesterol measured at baseline, 8th Week post treatment and 16th Week post treatment from intravenous blood specimen.
Change in Serum High Density Lipoprotein (HDL-C) | 16 Weeks
  Serum High Density Lipoprotein (HDL-C) measured at baseline, 8th Week post treatment and 16th Week post treatment from intravenous blood specimen.
Change in Serum High Density Lipoprotein (LDL-C) | 16 Weeks
  Serum High Density Lipoprotein (LDL-C) measured at baseline, 8th Week post treatment and 16th Week post treatment from intravenous blood specimen.
Change in Forced Expiratory Volume - 01 Second (FEV1) | 16 Weeks
  Forced Expiratory Volume - 01 Second (FEV1) measured at baseline, 8th Week post treatment and 16th Week post treatment using digital spirometer.
Change in Forced Expiratory Volume 1 Second / Forced Vital Capacity (FEV1/FVC) | 16 Weeks
  Forced Expiratory Volume 1 Second / Forced Vital Capacity (FEV1/FVC) measured at baseline, 8th Week post treatment and 16th Week post treatment using digital spirometer.
Change in Peak Expiratory Flow Rate (PEFR) | 16 Weeks
  Peak Expiratory Flow Rate (PEFR) measured at baseline, 8th Week post treatment and 16th Week post treatment using digital spirometer.
Change in Body Fat Percentage | 16 Weeks
  Body Fat Percentage measured at baseline, 8th Week post treatment and 16th Week post treatment using a body fat analyzer
Change in Waist-Hip Ratio | 16 Weeks
  Waist-Hip Ratio measured at baseline, 8th Week post treatment and 16th Week post treatment. Waist and hip circumference will be measured using inelastic tape.
Change in Hand Grip Strength | 16 Weeks
  Hand Grip Strength (Dominant & Non Dominant)measured at baseline, 8th Week post treatment and 16th Week post treatment using Hand Held Dynamometer.
Change in VO2 Maximum | 16 Weeks
  VO2 Maximum measured at baseline, 8th Week post treatment and 16th Week post treatment using treadmill.
Change in Level of Perceived Exertion | 16 Weeks
  Level of Perceived Exertion measured at baseline, 8th Week post treatment and 16th Week post treatment using BROG scale.

CONTACTS AND LOCATIONS:
Overall Officials: Danish Hassan, PhD*, Principal Investigator — Riphah International University; Syed Shakil ur Rehman, PhD, Study Director — Riphah International University
Locations (1):
- Riphah Rehabiliation Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] AlGhatrif M, Lakatta EG. The conundrum of arterial stiffness, elevated blood pressure, and aging. Curr Hypertens Rep. 2015 Feb;17(2):12. doi: 10.1007/s11906-014-0523-z. PMID 25687599
- [Background] Mills KT, Bundy JD, Kelly TN, Reed JE, Kearney PM, Reynolds K, Chen J, He J. Global Disparities of Hypertension Prevalence and Control: A Systematic Analysis of Population-Based Studies From 90 Countries. Circulation. 2016 Aug 9;134(6):441-50. doi: 10.1161/CIRCULATIONAHA.115.018912. PMID 27502908
- [Background] Park JB, Kario K, Wang JG. Systolic hypertension: an increasing clinical challenge in Asia. Hypertens Res. 2015 Apr;38(4):227-36. doi: 10.1038/hr.2014.169. Epub 2014 Dec 11. PMID 25503845
- [Background] Lee CJ, Kim JY, Shim E, Hong SH, Lee M, Jeon JY, Park S. The Effects of Diet Alone or in Combination with Exercise in Patients with Prehypertension and Hypertension: a Randomized Controlled Trial. Korean Circ J. 2018 Jul;48(7):637-651. doi: 10.4070/kcj.2017.0349. PMID 29968437
- [Background] Gerber M, Beck J, Brand S, Cody R, Donath L, Eckert A, Faude O, Fischer X, Hatzinger M, Holsboer-Trachsler E, Imboden C, Lang U, Mans S, Mikoteit T, Oswald A, Puhse U, Rey S, Schreiner AK, Schweinfurth N, Spitzer U, Zahner L. The impact of lifestyle Physical Activity Counselling in IN-PATients with major depressive disorders on physical activity, cardiorespiratory fitness, depression, and cardiovascular health risk markers: study protocol for a randomized controlled trial. Trials. 2019 Jun 20;20(1):367. doi: 10.1186/s13063-019-3468-3. PMID 31221205
- [Background] Zheng S, Lubin B, Au R, Murabito JM, Benjamin EJ, Shwartz M. Advantages of Continuous-Valued Risk Scores for Predicting Long-Term Costs: The Framingham Coronary Heart Disease 10-Year Risk Score. Adv Geriatr Med Res. 2019;1(1):e190004. doi: 10.20900/agmr20190004. Epub 2019 Jun 6. PMID 31448373
- [Background] Zhang C, Zhang Y, Lin H, Liu S, Xie J, Tang Y, Huang H, Zhang W. Blood pressure control in hypertensive patients and its relation with exercise and exercise-related behaviors: A case-control study. Medicine (Baltimore). 2020 Feb;99(8):e19269. doi: 10.1097/MD.0000000000019269. PMID 32080136